CLINICAL TRIAL: NCT03230162
Title: Sildenafil Versus Low Molecular Weight Heparin in Fetal Growth Restriction Treatment
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Radwa Rasheedy Ali, lecturer of obstetrics and gynecology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ain shams university maternity
Record Dates: First submitted 2017-05-28; First posted 2017-07-26 (Actual); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Fetal Growth Abnormality; Fetal Growth Restriction
MeSH Terms: conditions — Fetal Growth Retardation | interventions — Sildenafil Citrate; Heparin, Low-Molecular-Weight; Tinzaparin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sildenafil citrate (Experimental): 50 pregnant female will be treated with sildenafil citrate 25 mg every 8 hours (Silden EIPICO co.) orally, starting at the diagnosis of FGR till delivery.
  Interventions: Drug: Sildenafil
- low molecular weight heparin (Experimental): 50 pregnant female will be treated with a single daily dose of LMWH (tinzaparin) (Innohep LEO pharmaceutical products.) subcutaneously starting at diagnosis of FGR till delivery according to body weight as follow < 50 kg 3500 units daily 50-90 kg 4500 units daily 91-130 kg 7000 units daily 131-170 kg 9000 units daily > 170 kg 75 u/kg/day
  Interventions: Drug: low molecular weight heparin

INTERVENTIONS:
Drug: Sildenafil — sildenafil citrate 25 mg every 8 hours (Silden EIPICO co.) orally, starting at the diagnosis of FGR till delivery
  Other Names: Silden EIPICO co.
  Arms: sildenafil citrate
Drug: low molecular weight heparin — a single daily dose of LMWH (tinzaparin) (Innohep LEO pharmaceutical products.) subcutaneously starting at diagnosis of FGR till delivery
  Other Names: tinzaparin; Innohep LEO pharmaceutical products
  Arms: low molecular weight heparin

SUMMARY:
comparing the effect of using sildenafil citrate and LMWH in treatment of cases of IUGR due to placental insufficiency

DETAILED DESCRIPTION:
One hundred pregnant women with documented intrauterine growth restriction due to placental insufficiency at 28-35 weeks of gestation will be distributed into two groups:

* Group S: 50 women will receive Sildenafil citrate 25 mg tab 3 times daily.
* Group H: 50 women will receive single dose of LMWH subcutaneous daily.

Both groups will undergo strict fetal surveillance in the form of:

Umbilical artery Doppler (UAD) is the primary surveillance tool in the FGR fetus:

middle cerebral artery (MCA) Doppler, ultrasound for (AC, EFW, and deepest vertical pocket (DVP) for amniotic fluid) and non stress test and Biophysical profile (BPP)

ELIGIBILITY:
Inclusion Criteria:

* Maternal age between 20-35 years.
* Being at a gestational age 28-35wks.
* Singleton pregnancy.
* Fetal growth restriction diagnosed by ultrasound with estimated fetal weight below the 10th percentile, and/or fetal abdominal circumference at or below the tenth percentile.

Exclusion Criteria:

* Maternal age less than 20 years or more than 35 years.
* Undetermined gestational age.
* Multiple gestation.
* Chronic diseases with pregnancy e.g. Chronic hypertension, diabetes type 1 or 2.
* Etiologies of FGR other than placental insufficiency as fetal malformations, aneuploidy or infections.
* Suspected fetal compromise requiring emergency delivery.
* Any contraindication to the use of sildenafil e.g. known significant maternal cardiac disease, left ventricular outflow tract obstruction, concomitant treatment with nitrates or previous allergy to sildenafil.
* Any contraindication to the use of LMWH e.g. known bleeding disorder, active antenatal bleeding or at increased risk of major hemorrhage (e.g. placenta praevia), thrombocytopenia, severe renal or hepatic disease.
* Drug or alcohol abuse.
* Patient refusing to participate in the study or unable to consent.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-05-01 (Estimated); Study Completion 2018-05-01 (Estimated)

PRIMARY OUTCOMES:
Neonatal birth weight in grams | At time of Delivery

SECONDARY OUTCOMES:
The change in Doppler velocity indices, | 24 week till 35 weeks
Fetal growth velocity | weekly till time of delivery
Gestational age at delivery, | at time of delivery
APGAR score | at 1 and 5 min of life
Neonatal complication rates | The first 28 day of delivery
  respiratory distress syndrome, intraventricular hemorrhage (IVH), neonatal necrotizing enterocolitis (NEC), neonatal anemia, and neonatal blood transfusion
Neonatal ICU admission rate | The first 28 day of delivery
the interval between the diagnosis and delivery | at time of delivery

CONTACTS AND LOCATIONS:
Locations (1):
- AinShams university maternity hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided